CLINICAL TRIAL: NCT05410080
Title: the Efficacy of Fetal Arterial and Venous Doppler Indices in Predicting Perinatal Outcome Among Diabetic Pregnant Patients
Brief Title: the Efficacy of Fetal Arterial and Venous Doppler Indices in Predicting Perinatal Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany saad, assistant professor, Cairo University
Other Study IDs: Hany Saad
Record Dates: First submitted 2022-05-06; First posted 2022-06-08 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Gestational Diabetes; Pre-Gestational Diabetes; IUGR; Macrosomia, Fetal
MeSH Terms: conditions — Diabetes, Gestational; Fetal Macrosomia | interventions — Postprandial Period; Echocardiography, Doppler

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- good perinatal outcome: Fasting blood sugar 2 hours postprandial HBA1C Ultrasound and Doppler
  Interventions: Diagnostic Test: Fasting blood sugar, 2 hours postprandial, HBA1C ,Ultrasound and Doppler study
- poor perinatal outcome: Fasting blood sugar 2 hours postprandial HBA1C Ultrasound and Doppler
  Interventions: Diagnostic Test: Fasting blood sugar, 2 hours postprandial, HBA1C ,Ultrasound and Doppler study

INTERVENTIONS:
Diagnostic Test: Fasting blood sugar, 2 hours postprandial, HBA1C ,Ultrasound and Doppler study — Fasting blood sugar, 2 hours postprandial, HBA1C ,Ultrasound and Doppler study

SUMMARY:
To determine and evaluate the diagnostic performance of Doppler sonography of umbilical artery (UA), fetal middle cereberal artery (MCA), ductus venosus (VD) and umbilical vein (UV) for prediction of adverse perinatal outcome among diabetic pregnant women.

DETAILED DESCRIPTION:
The included women age will range between 18 and 35 years old. They will be pregnant in a singleton healthy living fetus at a gestational age between 34 and 39 weeks (confirmed by a reliable date for the last menstrual period or/and 1st trimester ultrasound scan). Women with other maternal medical disorders that may affect perinatal outcome rather than diabetes will be excluded from the study. Exclusion criteria also include women with pre-labour rupture of membrane, antepartum hemorrhage, fetuses with congenital anomalies and those who will receive respiratory depressants (e.g., opioid analgesics) within 2 hours of delivery. According to NICE guidelines 2015[13], gestational diabetes is diagnosed if the woman has either:

* A fasting plasma glucose level of 5.6 mmol/litre (100 mg/dL) or above Or
* A 2-hour plasma glucose level of 7.8 mmol/litre (140 mg/dL) or above. Informed written consents will be obtained from all participants after explanation of the study and its aims. All participants be subjected to the following: Full history taking [including a detailed history of the diabetes state during the current pregnancy [e.g., onset, course, duration, type, current medications and whether the blood sugar level is controlled or not ], complete physical examination including general [ BMI & blood pressure measurement] and obstetric examinations, laboratory investigations [Complete blood count - fasting blood sugar,2 hours postprandial & HBA1C - liver enzymes & kidney function-urine analysis for glucosuria and ketonuria] and obstetric ultrasound [to confirm fetal viability & number, to assess gestational age, estimated fetal weight, and growth percentile and to measure amniotic fluid index] and fetal Doppler ultrasonography assessment using GE Voluson Pro-V and GE Voluson E10 (GE Healthcare, Milwaukee, WI, USA) ultrasonography system with 3.5-5 MHz abdominal transducer. The color flow imaging (to identify the vessels) & pulsed wave velocimetry will be used to obtain flow velocity waveforms within 24 hours of pregnancy termination. In all Doppler studies, while the woman is lying in a semi-recumbent position, the angle of insonation of the vessels is less than 45 degrees; the high-pass filter is set at 100 Hz. Care is taken not to exert undue pressure on the fetal head because this alters the flow velocity waveforms from the MCA. Furthermore, examination of the fetal vessels will be performed in the absence of fetal body and respiratory movements, with a fetal heart rate ranging from 120-160 beats per minute. Measurements will be obtained from ≥ 4 consecutive flow velocity waveforms of good quality and averaged. Umbilical artery (UA) Doppler will be evaluated from a free- floating loop in the mid portion of the cord. Middle cerebral artery (MCA) Doppler will be obtained from a transverse image of the fetal head at the level of sphenoid bones.

Colour flow imaging will be used to display the circle of Willis. Then, calculation of the cerebro-placental ratio (CPR) will be done. Ductus venosus (DV) Doppler will be sampled soon after its origin from the umbilical vein. Also measurement of fetal umbilical vein (UV) flow will be done.

From the flow velocity waveforms of the UA and MCA, the pulsatility index (PI) & the resistance index (RI) will be measured. From the flow velocity waveforms of the DV, peak velocity index (PVIV), peak systolic velocity (PSV) and A wave will be measured.

From the umbilical vein flow, the presence or absence of pulsatile flow will be recorded.

All labours will be attended by an expert neonatologist who will be blinded to the results of Doppler indices measurements & the following will be recorded: APGAR score at (1 & 5 min) -Neonatal birth weight - Fetal growth restriction (FGR) will be defined as birth weight of less than 10 th percentile of newborn weight in normal pregnancies at corresponding gestational age - Fetal macrosomia will be defined as birth weight of more than 90th percentile of newborn weight in normal pregnancies at corresponding gestational age - The occurrence of respiratory complications [Transient Tachypnea of the newborn (TTN) or Respiratory Distress Syndrome (RDS)] - The occurrence of neonatal hypoglycemia was defined as blood glucose level less than 2 mmol/liter (35 mg/dL) - The further need for neonatal intensive care unit (NICU) admission and Perinatal death.

ELIGIBILITY:
Inclusion Criteria:

* The included women age will range between 18 and 35 years old.
* They will carry a singleton healthy living fetus at a gestational age between 34 and 39 weeks (confirmed by a reliable date for the last menstrual period or/and 1st trimester ultrasound scan).
* known to be diabetic in the current pregnancy (PGDM or GDM).

Exclusion Criteria:

* Women with other maternal medical disorders that may affect perinatal outcome rather than diabetes were excluded from the study.
* women with pre-labour rupture of membrane.
* antepartum hemorrhage, fetuses with congenital anomalies .
* who will receive respiratory depressants (e.g., opioid analgesics) within 2 hours of delivery.

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — pregnant female
Study Population: 140 pregnant women, will be recruited from emergency and inpatients departments.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-09-20 (Estimated); Study Completion 2022-10-20 (Estimated)

PRIMARY OUTCOMES:
The diagnostic value of umbilical artery (UA) Doppler indices in predicting adverse perinatal outcome among diabetic pregnant patients | within 24 hours before delivery
  The diagnostic value of umbilical artery (UA) Doppler indices (RI & PI) in predicting adverse perinatal outcome among diabetic pregnant patients.
  Sensitivity and specificity of umbilical artery RI & PI in detecting adverse perinatal outcome.
The diagnostic value of middle cerebral artery (MCA) Doppler indices in predicting adverse perinatal outcome among diabetic pregnant patients | within 24 hours before delivery
  The diagnostic value of middle cerebral artery (MCA) Doppler indices (RI & PI) in predicting adverse perinatal outcome among diabetic pregnant patients.
  Sensitivity and specificity of middle cerebral artery RI & PI in detecting adverse perinatal outcome.

SECONDARY OUTCOMES:
The diagnostic value of cerebroplacental ratio (CPR) in predicting adverse perinatal outcome among diabetic pregnant patients. | within 24 hours before delivery
  The diagnostic value of cerebroplacental ratio (CPR) [MCA/UA PI] in predicting adverse perinatal outcome among diabetic pregnant patients.
  Sensitivity and specificity of CPR in detecting adverse perinatal outcome.
The diagnostic value of ductus venosus Doppler indices in predicting adverse perinatal outcome among diabetic pregnant patients. | within 24 hours before delivery
  The diagnostic value of ductus venosus Doppler indices ( PVIV,PSV and abnormal A wave) in predicting adverse perinatal outcome among diabetic pregnant patients.
  Sensitivity and specificity of ductus venosus PVIV,PSV and abnormal A wave in detecting adverse perinatal outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hany Saad, MD, Principal Investigator — Kasr Alainy Hospital(Faculty of Medicine -Cairo university
Locations (2):
- Egypt (2):
  - Cairo University, Cairo
  - Kasr Alainy hospital (Faculty of Medicine-Cairo University), Cairo